CLINICAL TRIAL: NCT03297372
Title: Clinical Study to Investigate Visual Performance of Hydrophobic Monofocal IOL: MicroPure 1.2.3.
Brief Title: Visual Performance Intraocular Lens (IOL) MicroPure 1.2.3.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY1604
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Cataract; Lens Opacities
Keywords: Intraocular lens; monofocal; cataract; PhysIOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IOL Implantation experimental (Experimental): Implantation of Micropure 1.2.3. in one of the eyes of the study subject
  Interventions: Device: IOL implantation

INTERVENTIONS:
Device: IOL implantation — Implantation of monofocal IOL Micropure 1.2.3

SUMMARY:
The clinical investigation is a post-market clinical follow up study whereby patients undergoing routine cataract surgery will have monolateral implantation of a commercially available, CE approved monofocal intraocular lens MicroPure 1.2.3. (PhysIOL, Liège, Belgium).

DETAILED DESCRIPTION:
The examinations consist of visual acuity data, contrast sensitivity exams, slitlamp examinations and posterior capsule opacification (PCO) grading.

Follow up will be up to 24 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent

Exclusion Criteria:

* Irregular astigmatism
* Age of patient < 45 years
* Regular corneal astigmatism > 0.75 D on study eye as measured by an automatic keratometer (regularity determined by the topography of the keratometry)
* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* Complicated surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
monocular Corrected Distance Visual Acuity (CDVA) under photopic conditions | 6 months postoperative
  The primary study end point is to show statistically equal visual acuity outcomes on monocular Corrected Distance Visual Acuity (CDVA) under photopic conditions compared to literature data on a monofocal hydrophobic IOL (Alcon - Acrysof SN60AT).

SECONDARY OUTCOMES:
Posterior capsule opacification (PCO) grading | 2 years postoperative
  grade of the PCO determined by slitlamp
Uncorrected Distance Visual acuity (UDVA) | 6 months postoperative
  Monocular Uncorrected Distance Visual acuity (UDVA)
Contrast Sensitivity | 6 months postoperative
  Contrast Sensitivity under photopic and mesopic light conditions
Glistening assessment | 2 years postoperative
  Assessment of glistenings by slitlamp determination

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Schiano, MD, Principal Investigator — Fondazione GB Bietti - IRCCS
Locations (2):
- Italy (2):
  - Azienda Ospedaliera San Giovanni Addolorata - presidio Britannico, Rome
  - Fondazione GB Bietti - IRCCS, Rome

IPD SHARING:
Plan to Share IPD: No